CLINICAL TRIAL: NCT07373132
Title: Effects of Aromatherapy on Sleep Quality in Hospitalized Elderly Female Patients With Insomnia: Protocol for A Randomized, Double-Blind, Placebo-Controlled Parallel Trial
Brief Title: Effects of Aromatherapy on Sleep Quality in Hospitalized Elderly Female Patients With Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Zengzeng Wei, Clinical Professor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZWei
Record Dates: First submitted 2026-01-10; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to receive either standardized aromatherapy (lavender essential oil) or placebo (odorless fractionated coconut oil) for five consecutive nights
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aromatherapy (Experimental)
  Interventions: Other: Aromatherapy
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — Verify patient identity and explain the intervention. Ensure comfortable supine or semi-recumbent position. Drop 2 drops of lavender essential oil onto a sterile cotton ball; place inside disposable urine cup.
  Position cup 20 cm from patient's nostrils; instruct patient to perform 10 deep breaths.
  Place cup at bedside until morning. Lay treatment cloth under patient's wrists. Apply 1 drop of lavender oil to both thumbs, perform bilateral Shenmen (HT7) acupoint pressure on the wrist Shenmen acupoint pressure for 10 minutes per side, moderate pressure causing mild local distension but no pain.
  Restore patient to comfortable position; remove materials; wash hands. Record any immediate reactions or discomfort.
  Arms: aromatherapy
Other: Placebo — Identical procedure using odorless fractionated coconut oil. Sham acupoint pressure on a non-acupoint location near the wrist performed identically to maintain blinding.
  Arms: placebo

SUMMARY:
To evaluate the efficacy and safety of standardized aromatherapy compared with placebo in improving sleep quality among hospitalized elderly female patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥60 years.
* Hospitalized in the Second Affiliated Hospital of Anhui Medical University.
* Athens Insomnia Scale (AIS) >6.
* Ability to communicate and understand instructions.
* Non-allergic to essential oils.
* Fully informed and voluntarily consent to participate.

Exclusion Criteria:

* Cognitive impairment-.
* History of hypersensitivity to aromatherapy oils.
* Use of sedative-hypnotic medications within past 2 weeks.
* Sleep disorders secondary to organic or psychiatric diseases.
* Unable to comply with study procedures.

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Athens Insomnia Scale | Evaluated at baseline, day 6 and 2-week follow-up.
  Total score 0-24; higher scores indicate worse insomnia.